CLINICAL TRIAL: NCT00338143
Title: A Phase IIIb, Open-Label, Multicenter Study to Evaluate the Safety of 1.0 mg/kg Subcutaneously Administered Efalizumab in Adults With Moderate to Severe Plaque Psoriasis, Including Those Who Are Receiving Concomitant Antipsoriatic Therapies or Have Recently Transitioned From Systemic Therapies
Brief Title: A Study to Evaluate Efalizumab in Adults With Plaque Psoriasis, Including Those Who Are Receiving Concomitant Antipsoriatic Therapies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACD2782g
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: Psoriasis
Keywords: Plaque psoriasis; Antipsoriatic
MeSH Terms: conditions — Psoriasis | interventions — efalizumab

INTERVENTIONS:
Drug: efalizumab

SUMMARY:
This is a Phase IIIb, open label, uncontrolled, multicenter study designed to evaluate the safety and tolerability of 12 weeks of subcutaneously administered efalizumab in subjects with moderate to severe plaque psoriasis who are candidates for systemic therapy and may also be receiving topical therapies, PUVA, or UVB phototherapy during the efalizumab treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Plaque psoriasis covering >=10% of total BSA
* Plaque psoriasis diagnosed for at least 6 months
* In the opinion of the investigator, a candidate for systemic therapy for psoriasis
* 18-75 years old
* Body weight <=125 kg
* For women of childbearing potential, use of an acceptable method of contraception to prevent pregnancy and agreement to continue to practice an acceptable method of contraception for the duration of their participation in the study and for 3 months after the last dose of efalizumab

Exclusion Criteria:

* Guttate, erythrodermic, or pustular psoriasis as sole or predominant form of psoriasis
* Pregnancy or lactation
* Clinically significant psoriasis flare during screening or at the time of enrollment
* History of or ongoing uncontrolled bacterial, viral, fungal, or atypical mycobacterial infection
* History of opportunistic infections (e.g., systemic fungal infections, parasites)
* Seropositivity for hepatitis B or C virus
* Seropositivity for human immunodeficiency virus (HIV)
* History of active tuberculosis (TB) or currently undergoing treatment for TB
* Presence or history of malignancy within the past 5 years, including lymphoproliferative disorders
* Previous treatment with efalizumab (anti-CD11a)
* Diagnosis of hepatic cirrhosis, regardless of cause or severity
* Hospital admission for cardiovascular or pulmonary disease within the last year
* History of severe allergic or anaphylactic reactions to monoclonal antibodies or fusion proteins, which contain an Ig Fc region (e.g., etanercept, alefacept)
* History of treatment with lymphocyte-depleting monoclonal antibodies or immunoadhesion molecules (e.g., anti-CD4, CTLA4-Ig, alefacept)
* White blood cell (WBC) count < 4000/uL or > 14,000/uL
* Hepatic enzymes >= 3 times the upper limit of normal
* Creatinine >= 2 times the upper limit of normal
* Use of experimental drugs or treatments within 30 days or five half-lives, whichever is longer, prior to the first dose of efalizumab
* Use of a live virus or live bacteria vaccine in the 14 days prior to the first dose of efalizumab
* Any medical condition that, in the judgment of the investigator, would jeopardize the subject's safety following exposure to study drug or would significantly interfere with the subject's ability to comply with the provisions of this protocol
* Restrictions and/or directions apply to the following treatments during specified time periods prior to and during the efalizumab treatment period: Systemic therapy for psoriasis (biologic and non-biologic); Systemic immunosuppressive drugs for conditions other than psoriasis; Live virus or bacteria vaccine (these vaccines may include, but are not limited to, measles, mumps, rubella, polio, BCG, yellow fever, and TY21a typhoid); Other vaccines or allergy desensitization injections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200
Dates: Start 2003-10; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivor Caro, M.D., Study Director — Genentech, Inc.